CLINICAL TRIAL: NCT00087438
Title: A Phase II Trial of Stereotactic Body Radiation Therapy (SBRT) in the Treatment of Patients With Medically Inoperable Stage I/II Non-Small Cell Lung Cancer
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Inoperable Stage I or Stage II Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0236; CDR0000371578
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2018-12

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic body radiation therapy (SBRT) (Experimental): 20 Gy per fraction for 3 fractions over 1.5-2 weeks, for a total of 60 Gy
  Interventions: Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Stereotactic body radiation therapy may be able to deliver x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying how well stereotactic body radiation therapy works in treating patients with inoperable stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether treatment with stereotactic body radiotherapy results in acceptable local control (i.e., ≥ 80%) in patients with medically inoperable stage I or II non-small cell lung cancer.

Secondary

* Determine treatment-related toxicity in patients treated with this therapy.
* Determine disease-free survival, overall survival, and patterns of failure in patients treated with this therapy.

OUTLINE: This is a multicenter study.

Patients receive 3 fractions of stereotactic body radiotherapy over 8-14 days in the absence of disease progression or unacceptable toxicity.

Patients are followed up at 6 and 12 weeks, every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study within 26 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * The following primary cancer subtypes are eligible:

    * Squamous cell carcinoma
    * Adenocarcinoma
    * Large cell carcinoma
    * Bronchoalveolar cell carcinoma
    * Non-small cell carcinoma not otherwise specified
* Stage I or II disease based on 1 of the following tumor node metastasis (TNM) stage criteria:

  * T1, N0, M0
  * T2 (≤ 5 cm), N0, M0
  * T3 (≤ 5 cm), N0, M0 (chest wall primary tumors only)
* No primary tumor of any T-stage within or touching the zone of the proximal bronchial tree* NOTE: *Defined as a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, and right and left lower lobe bronchi)
* No primary T3 tumors involving the central chest (≤ 2 cm toward carina invasion) or structures of the mediastinum
* Any hilar or mediastinal lymph nodes > 1 cm on CT scan OR demonstrating suspicious uptake on positron-emission tomography scan must be biopsied and confirmed negative for NSCLC
* The primary tumor must be deemed technically resectable with a reasonable possibility of obtaining a gross total resection with negative margins (defined as a potentially curative resection (PCR))
* Deemed medically inoperable based on pulmonary function for surgical resection of NSCLC secondary to an underlying physiological problem, including any of the following medical conditions*:

  * Baseline forced expiratory volume (FEV)_1< 40% of predicted
  * Postoperative predicted FEV_1 < 30% of predicted
  * Severely reduced diffusion capacity
  * Baseline hypoxemia and/or hypercapnia
  * Exercise oxygen consumption < 50% of predicted
  * Severe pulmonary hypertension
  * Diabetes mellitus with severe end organ damage
  * Severe cerebral, cardiac, or peripheral vascular disease
  * Severe chronic heart disease NOTE: *Patients who refuse a PCR due to preference, ideology, emotional or psychological issues, mental illness, or inability to give informed consent are not eligible
* No evidence of regional or distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* See Disease Characteristics
* No active pericardial infection

Pulmonary

* See Disease Characteristics
* No active pulmonary infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active systemic infection
* No other concurrent illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy
* No concurrent vaccine therapy

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior lung or mediastinal radiotherapy
* No concurrent standard fractionated radiotherapy
* No concurrent intensity modulated radiotherapy
* No concurrent cobalt-60 or charged particle beams (including electrons, protons, or heavier ions)

Surgery

* See Disease Characteristics
* No concurrent surgery

Other

* No other concurrent antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-05; Primary Completion 2010-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Principal Investigator — Simmons Cancer Center
Locations (2):
- United States (2):
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Background] Hurkmans CW, Cuijpers JP, Lagerwaard FJ, Widder J, van der Heide UA, Schuring D, Senan S. Dosimetric evaluation of heterogeneity corrections for RTOG 0236: stereotactic body radiotherapy of inoperable Stage I-II non-small-cell lung cancer. In reply to Dr. Xiao et al. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):318; author reply 318. doi: 10.1016/j.ijrobp.2009.05.050. No abstract available. PMID 19695451
- [Background] Timmerman R, Galvin J, Michalski J, Straube W, Ibbott G, Martin E, Abdulrahman R, Swann S, Fowler J, Choy H. Accreditation and quality assurance for Radiation Therapy Oncology Group: Multicenter clinical trials using Stereotactic Body Radiation Therapy in lung cancer. Acta Oncol. 2006;45(7):779-86. doi: 10.1080/02841860600902213. PMID 16982540
- [Result] Timmerman R, Paulus R, Galvin J, Michalski J, Straube W, Bradley J, Fakiris A, Bezjak A, Videtic G, Johnstone D, Fowler J, Gore E, Choy H. Stereotactic body radiation therapy for inoperable early stage lung cancer. JAMA. 2010 Mar 17;303(11):1070-6. doi: 10.1001/jama.2010.261. PMID 20233825
- [Result] Xiao Y, Papiez L, Paulus R, Timmerman R, Straube WL, Bosch WR, Michalski J, Galvin JM. Dosimetric evaluation of heterogeneity corrections for RTOG 0236: stereotactic body radiotherapy of inoperable stage I-II non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2009 Mar 15;73(4):1235-42. doi: 10.1016/j.ijrobp.2008.11.019. PMID 19251095
- [Result] Timmerman RD, Paulus R, Galvin J, et al.: Toxicity analysis of RTOG 0236 using stereotactic body radiation therapy to treat medically inoperable early stage lung cancer patients. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-151, S86, 2007.

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiation Therapy (SBRT): 20 Gy per fraction for 3 fractions over 1.5-2 weeks, for a total of 60 Gy
  stereotactic body radiation therapy
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Started | 59
Completed | 55 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 4
Not completed — Ineligible / No protocol treatment | 4

BASELINE CHARACTERISTICS:
Population: All eligible patients who received protocol treatment.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 72 [48 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Local Control at 2 Years
Description: Local control is defined as absence of local failure, which is defined as the combination of primary tumor failure (PTF) or involved lobe failure (ILF). PTF was defined based on meeting two criteria: 1. Local enlargement defined as ≥ 20% increase in the longest diameter of the gross tumor volume (GTV) per computerized tomography (CT), and 2. Evidence of tumor viability. Tumor viability could be affirmed by either demonstrating positron emission tomography (PET) imaging with uptake of a similar intensity as the pretreatment staging PET, or by repeat biopsy confirming carcinoma. PTF included marginal failures occurring within 1 cm of the planning target volume (PTV). ILF is defined as failure beyond the primary tumor but within the involved lobe. Local control time is defined as time from start of treatment to the the date of local recurrence, last known follow-up (censored), or death without local failure (censored). Rates are estimated using the Kaplan-Meier method.
Time Frame: From the start of treatment to 2 years
Population: Eligible patients who started protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
percentage of subjects | 97.6 [84.3 to 99.7]
Statistical Analysis 1: Comparison: Stereotactic Body Radiation Therapy (SBRT); Null hypothesis = 60% two-year local control (0.02128/mo. hazard rate); alternative = 80% (0.0093/mo.) assuming at least approximately exponential distribution of time to local progression. Using the asymptotic properties of the ratio of the logarithms of hazard rates, less than 18 cases of local progression were required for a Type I error rate of 0.05 with 80% power to detect a difference in local control rates at least this large. Hazard rate estimated using life table two-year estimates; Test type: Superiority or Other; p = 0.013, z-test, one-sided — Test statistic = [ln(estimated hazard rate) - ln(hypothesized hazard rates)] / [1/square root (number of patients with local progression by two years]. Reject null hypothesis at an alpha level of 0.05 if test statistics is less than -1.645

2. Secondary Outcome: Proportion of Subjects With Specified Adverse Events
Description: Specified adverse events are defined as any treatment-related adverse events that are grade 4, grade 5, or any of the following treatment-related grade 3 adverse events:
  * Gastrointestinal: dysphagia, esophagitis, esophageal stricture, esophageal ulceration;
  * Cardiac: pericarditis, pericardial effusion, cardiomyopathy, ventricular dysfunction;
  * Neurologic: myelitis, neuropathy (cranial and motor)
  * Hemorrhage: pulmonary or upper respiratory
  * Pulmonary: decline in pulmonary function as measured by pulmonary function tests, pneumonitis, pulmonary fibrosis, hypoxemia, pleural effusion.
  Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The Common Terminology Criteria for Adverse Events (CTCAE) v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From randomization to last follow-up. Analysis occurred after all patients had been on study for at least 2 years. Maximum follow-up at time of analysis was 4.2 years.
Population: All eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
Participants | 9

3. Secondary Outcome: Rate of Local Recurrence at 2 Years
Description: Local failure is defined as the combination of primary tumor failure (PTF) or involved lobe failure (ILF). PTF was defined based on meeting two criteria: 1. Local enlargement defined as ≥ 20% increase in the longest diameter of the gross tumor volume (GTV) per computerized tomography (CT), and 2. Evidence of tumor viability. Tumor viability could be affirmed by either demonstrating positron emission tomography (PET) imaging with uptake of a similar intensity as the pretreatment staging PET, or by repeat biopsy confirming carcinoma. PTF included marginal failures occurring within 1 cm of the planning target volume (PTV). ILF is defined as failure beyond the primary tumor but within the involved lobe. Time to local recurrence is defined as time from start of treatment to the the date of local recurrence, last known follow-up (censored), or death without local recurrence (censored).
Time Frame: From the start of treatment to 2 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
percentage of participants | 2.4 [0.3 to 15.7]

4. Secondary Outcome: Rate of Regional Recurrence at 2 Years
Description: Regional recurrence is defined as hilar, mediastinal, and supraclavicular nodal failure.Time to regional recurrence is defined as time from start of treatment to the date of first regional recurrence, last known follow-up (censored), or death without regional recurrence (competing risk). Rates are estimated using the cumulative incidence method.
Time Frame: From the start of treatment to 2 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
percentage of participants | 0 [0 to 0]

5. Secondary Outcome: Rate of Disseminated Recurrence at 2 Years
Description: Disseminated recurrence is defined as uninvolved lobe failures and failures beyond the lungs and regional lymph nodes. Time to disseminated recurrence is defined as time from start of treatment to the the date of disseminated recurrence, last known follow-up (censored), or death without disseminated recurrence (competing risk). Rates are estimated using the cumulative incidence method.
Time Frame: From the start of treatment to 2 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
percentage of participants | 11.1 [5.1 to 23.0]

6. Secondary Outcome: Rate of Disease-free Survival at 2 Years
Description: Disease is defined as local or regional progression or development of distant metastases. Disease-free survival time is defined as time from start of treatment to the date of disease, death, or last known follow-up (censored). Disease-free survival rates are estimated using the Kaplan-Meier method.
Time Frame: From the start of treatment to 2 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
percentage of participants | 67.3 [53.2 to 78.0]

7. Secondary Outcome: Rate of Overall Survival at 2 Years
Description: Overall survival time is defined as time from start of treatment to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From the start of treatment to 2 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 55
percentage of participants | 72.7 [58.9 to 82.6]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Serious Adverse Events (participants affected / at risk) | 11/55
Other Adverse Events (participants affected / at risk) | 49/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiation Therapy (SBRT) (N=55)
Lymphatics - Other (Blood and lymphatic system disorders) | 1
Cardiac general - Other (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 8
Forced expiratory volume (Investigations) | 1
Metabolic/laboratory - Other (Investigations) | 1
Weight decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia NOS (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiation Therapy (SBRT) (N=55)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 6
Hemoglobin (Blood and lymphatic system disorders) | 13
Atrial fibrillation (Cardiac disorders) | 3
Abdominal pain NOS (Gastrointestinal disorders) | 4
Diarrhea NOS (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Vomiting NOS (Gastrointestinal disorders) | 5
Chest pain (General disorders) | 8
Edema: limb (General disorders) | 4
Fatigue (General disorders) | 21
Pain - Other (General disorders) | 3
Pyrexia (General disorders) | 3
Rigors (General disorders) | 3
Infection with Grade 3 or 4 neutrop (Infections and infestations) | 3
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 6
Fracture NOS (Injury, poisoning and procedural complications) | 9
Activated partial thromboplastin ti (Investigations) | 3
Blood alkaline phosphatase increase (Investigations) | 3
Blood bilirubin increased (Investigations) | 4
Blood creatinine increased (Investigations) | 6
Forced expiratory volume (Investigations) | 9
Lymphopenia (Investigations) | 5
Metabolic/laboratory - Other (Investigations) | 3
Pulmonary function test NOS decreas (Investigations) | 5
Weight decreased (Investigations) | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 9
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal/soft tissue - Other (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Renal/genitourinary - Other (Renal and urinary disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No